CLINICAL TRIAL: NCT00075673
Title: A Phase I Study of Weekly Administration of Oral Navelbine in Combination With the COX-2 Inhibitor Celebrex in Relapsed and/or Metastatic Breast Cancer
Brief Title: Vinorelbine and Celecoxib in Treating Women With Relapsed or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Paula Silverman, MD, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICC3102
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: celecoxib — Patients receive oral celecoxib twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Drug: vinorelbine ditartrate — Patients receive oral vinorelbine on days 7, 14, and 21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining vinorelbine with celecoxib may kill more tumor cells.

PURPOSE: Phase I trial to determine the effectiveness of combining vinorelbine with celecoxib in treating women who have relapsed or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of vinorelbine and celecoxib in women with relapsed or metastatic breast cancer.
* Determine the safety profile of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive oral celecoxib twice daily on days 1-21 and oral vinorelbine on days 7, 14, and 21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of celecoxib and vinorelbine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 12-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Recurrent or metastatic (stage IV) disease
  * Incurable disease
* Measurable or evaluable disease
* Stable brain metastases allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 8.0 g/dL

Hepatic

* Bilirubin normal
* AST/ALT ≤ 2.5 times upper limit of normal

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min
* No clinically significant proteinuria
* No impaired renal function

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina
* No cardiac arrhythmia
* No inadequately controlled hypertension

Gastrointestinal

* No disorder that would alter gastrointestinal motility or absorption
* No dysphagia
* Able to swallow tablets or capsules

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No hypersensitivity to celecoxib

  * No prior urticaria, asthma, or other allergic-type reaction after taking aspirin or other nonsteroidal anti-inflammatory drugs
* No allergy to sulfa
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No ongoing or active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior trastuzumab (Herceptin®) and recovered
* No concurrent hematopoietic growth factors

Chemotherapy

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior adjuvant or neoadjuvant chemotherapy allowed
* Prior chemotherapy for recurrent or metastatic disease allowed
* No prior vinorelbine

Endocrine therapy

* At least 2 weeks since prior hormonal therapy
* Prior adjuvant or neoadjuvant hormonal therapy allowed
* Prior hormonal therapy for recurrent or metastatic disease allowed

Radiotherapy

* At least 4 weeks since prior radiotherapy for metastatic disease
* Prior adjuvant radiotherapy allowed

Surgery

* Not specified

Other

* At least 3 weeks since prior investigational anticancer agents and recovered
* At least 1 week since prior cyclooxygenase-2 (COX-2) inhibitors, except celecoxib
* No concurrent administration of any of the following drugs:

  * Lithium
  * Fluconazole
  * Aluminum antacids
  * Magnesium antacids
* Concurrent H_2 blocking agents or proton pump inhibitors allowed for the treatment of dyspepsia or gastroesophageal reflux disease
* Concurrent bisphosphonates allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-11; Primary Completion 2004-09 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of vinorelbine and celecoxib in women with relapsed or metastatic breast cancer. | Courses (21 days) repeat every 21 days in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Paula Silverman, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States